CLINICAL TRIAL: NCT02737020
Title: Rhodiola Rosea in Adults With Attention Deficit/Hyperactivity Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 150425
Record Dates: First submitted 2016-03-09; First posted 2016-04-13 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: ADHD; Adults; Treatment; Rhodiola rosea
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rhodiola (Experimental): Rhodiola rosea 200mg up to four times a day for 28 days
  Interventions: Drug: Rhodiola
- Placebo (Placebo Comparator): Placebo pill manufactured to mimic Rhodiola rosea 200mg, up to four times a day for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rhodiola — Rhodiola rosea 200mg pill up to four times a day
  Other Names: Rhodiola rosea
  Arms: Rhodiola
Drug: Placebo — up to four times a day
  Other Names: pill manufactured to mimic Rhodiola rosea 200mg
  Arms: Placebo

SUMMARY:
This study evaluates the use of Rhodiola rosea in the treatment of Attention Deficit/Hyperactivity Disorder (ADHD) in adults. Half of participants will receive Rhodiola rosea, while the other half will receive placebo.

DETAILED DESCRIPTION:
Rhodiola rosea is an herbal medicine used for centuries in various medical conditions. Many randomized controlled trials have evaluated its usefulness in stress and fatigue. There were benefits in attention in some of these studies. Mild side effects and beneficial antioxidant properties make reasonable an assessment of its potential benefits in adults with ADHD. To our knowledge, Rhodiola rosea was never studied in ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, (DSM-5) diagnostic criteria for ADHD in Adults
* Intelligence Quotient (IQ) above 70
* Eligibility to Rhodiola rosea

Exclusion Criteria:

* clinical contraindication fro Rhodiola rosea -
* any unstable chronic illness without proper treatment (hypertension, heart, kidney or liver disease)
* any significant neurological disease (delirium, dementia, epilepsy, AIDS, head trauma, multiple sclerosis, stroke, etc)
* unstable psychiatric comorbidities requiring immediate treatment (risk of suicide, current Substance Use Disorder, etc.)
* pregnant, nursing or absence of reliable contraception
* current use of nicotine (<30 days)
* use of anticoagulants
* current use of any psychoactive drug (<30 days)
* prior use of stimulants
* current or lifetime psychosis- current or lifetime bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Change in Swanson, Nolan and Pelham Rating Scale - Version IV (SNAP-IV) adapted to adults | Change from baseline SNAP-IV at 4 weeks

SECONDARY OUTCOMES:
Change in Adult Self-Report Scale (ASRS) | Change from baseline ASRS at 4 weeks

OTHER OUTCOMES:
Change in Wechsler Scale digit subtest (WAIS-III) | Change from baseline WAIS-III at 4 weeks
Change in Stop Signal Task | Change from baseline Stop Signal Task at 4 weeks
Change in Barkley Side Effect Rating Scale (SERS) | Change from baseline SERS at 4 weeks
  Including Rhodiola rosea side effects
Change in Insomnia Severity Index (ISI) | Change from baseline ISI at 4 weeks
Change in Beck-II Depression Scale | Change from baseline Beck-II Depression Scale at 4 weeks
Change in Beck Anxiety Scale | Change from baseline Beck Anxiety Scale at 4 weeks
Change in Adult ADHD Quality of Life Questionnaire (AAQoL) | Change from baseline AAQoL at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Grevet, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Swanson JM, Kraemer HC, Hinshaw SP, Arnold LE, Conners CK, Abikoff HB, Clevenger W, Davies M, Elliott GR, Greenhill LL, Hechtman L, Hoza B, Jensen PS, March JS, Newcorn JH, Owens EB, Pelham WE, Schiller E, Severe JB, Simpson S, Vitiello B, Wells K, Wigal T, Wu M. Clinical relevance of the primary findings of the MTA: success rates based on severity of ADHD and ODD symptoms at the end of treatment. J Am Acad Child Adolesc Psychiatry. 2001 Feb;40(2):168-79. doi: 10.1097/00004583-200102000-00011. PMID 11211365
- [Background] Brod M, Johnston J, Able S, Swindle R. Validation of the adult attention-deficit/hyperactivity disorder quality-of-life Scale (AAQoL): a disease-specific quality-of-life measure. Qual Life Res. 2006 Feb;15(1):117-29. doi: 10.1007/s11136-005-8325-z. PMID 16411036
- [Background] Kessler RC, Adler L, Ames M, Demler O, Faraone S, Hiripi E, Howes MJ, Jin R, Secnik K, Spencer T, Ustun TB, Walters EE. The World Health Organization Adult ADHD Self-Report Scale (ASRS): a short screening scale for use in the general population. Psychol Med. 2005 Feb;35(2):245-56. doi: 10.1017/s0033291704002892. PMID 15841682
- [Background] Mackin RS, Horner MD. Relationship of the Wender Utah Rating Scale to objective measures of attention. Compr Psychiatry. 2005 Nov-Dec;46(6):468-71. doi: 10.1016/j.comppsych.2005.03.004. PMID 16275215
- [Background] Sonuga-Barke EJ, Coghill D, Wigal T, DeBacker M, Swanson J. Adverse reactions to methylphenidate treatment for attention-deficit/hyperactivity disorder: structure and associations with clinical characteristics and symptom control. J Child Adolesc Psychopharmacol. 2009 Dec;19(6):683-90. doi: 10.1089/cap.2009.0024. PMID 20035586
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Gomes-Oliveira MH, Gorenstein C, Lotufo Neto F, Andrade LH, Wang YP. Validation of the Brazilian Portuguese version of the Beck Depression Inventory-II in a community sample. Braz J Psychiatry. 2012 Dec;34(4):389-94. doi: 10.1016/j.rbp.2012.03.005. PMID 23429809
- [Background] Gorenstein C, Andrade L. Validation of a Portuguese version of the Beck Depression Inventory and the State-Trait Anxiety Inventory in Brazilian subjects. Braz J Med Biol Res. 1996 Apr;29(4):453-7. PMID 8736107
- [Background] Seixas M, Weiss M, Muller U. Systematic review of national and international guidelines on attention-deficit hyperactivity disorder. J Psychopharmacol. 2012 Jun;26(6):753-65. doi: 10.1177/0269881111412095. Epub 2011 Sep 24. PMID 21948938
- [Background] Meszaros A, Czobor P, Balint S, Komlosi S, Simon V, Bitter I. Pharmacotherapy of adult attention deficit hyperactivity disorder (ADHD): a meta-analysis. Int J Neuropsychopharmacol. 2009 Sep;12(8):1137-47. doi: 10.1017/S1461145709990198. Epub 2009 Jul 7. PMID 19580697
- [Background] Iovieno N, Dalton ED, Fava M, Mischoulon D. Second-tier natural antidepressants: review and critique. J Affect Disord. 2011 May;130(3):343-57. doi: 10.1016/j.jad.2010.06.010. Epub 2010 Jun 26. PMID 20579741
- [Background] Panossian A, Wikman G, Sarris J. Rosenroot (Rhodiola rosea): traditional use, chemical composition, pharmacology and clinical efficacy. Phytomedicine. 2010 Jun;17(7):481-93. doi: 10.1016/j.phymed.2010.02.002. Epub 2010 Apr 7. PMID 20378318
- [Background] Hung SK, Perry R, Ernst E. The effectiveness and efficacy of Rhodiola rosea L.: a systematic review of randomized clinical trials. Phytomedicine. 2011 Feb 15;18(4):235-44. doi: 10.1016/j.phymed.2010.08.014. Epub 2010 Oct 30. PMID 21036578
- [Background] Darbinyan V, Kteyan A, Panossian A, Gabrielian E, Wikman G, Wagner H. Rhodiola rosea in stress induced fatigue--a double blind cross-over study of a standardized extract SHR-5 with a repeated low-dose regimen on the mental performance of healthy physicians during night duty. Phytomedicine. 2000 Oct;7(5):365-71. doi: 10.1016/S0944-7113(00)80055-0. PMID 11081987
- [Background] De Bock K, Eijnde BO, Ramaekers M, Hespel P. Acute Rhodiola rosea intake can improve endurance exercise performance. Int J Sport Nutr Exerc Metab. 2004 Jun;14(3):298-307. doi: 10.1123/ijsnem.14.3.298. PMID 15256690
- [Background] Shevtsov VA, Zholus BI, Shervarly VI, Vol'skij VB, Korovin YP, Khristich MP, Roslyakova NA, Wikman G. A randomized trial of two different doses of a SHR-5 Rhodiola rosea extract versus placebo and control of capacity for mental work. Phytomedicine. 2003 Mar;10(2-3):95-105. doi: 10.1078/094471103321659780. PMID 12725561
- [Background] Spasov AA, Wikman GK, Mandrikov VB, Mironova IA, Neumoin VV. A double-blind, placebo-controlled pilot study of the stimulating and adaptogenic effect of Rhodiola rosea SHR-5 extract on the fatigue of students caused by stress during an examination period with a repeated low-dose regimen. Phytomedicine. 2000 Apr;7(2):85-9. doi: 10.1016/S0944-7113(00)80078-1. PMID 10839209
- [Background] Olsson EM, von Scheele B, Panossian AG. A randomised, double-blind, placebo-controlled, parallel-group study of the standardised extract shr-5 of the roots of Rhodiola rosea in the treatment of subjects with stress-related fatigue. Planta Med. 2009 Feb;75(2):105-12. doi: 10.1055/s-0028-1088346. Epub 2008 Nov 18. PMID 19016404
- [Background] Logan GD, Cowan WB, Davis KA. On the ability to inhibit simple and choice reaction time responses: a model and a method. J Exp Psychol Hum Percept Perform. 1984 Apr;10(2):276-91. doi: 10.1037//0096-1523.10.2.276. PMID 6232345